CLINICAL TRIAL: NCT03433742
Title: Metal Ion Levels in Stryker Trident II Tritanium System with MDM Liner, Ceramic Head, and SecurFit Advanced Stems
Brief Title: Metal Ion Levels in Stryker Trident II Tritanium System with Modular Dual Mobility (MDM) Liner, Ceramic Head, and SecurFit Advanced Stems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-1567
Record Dates: First submitted 2018-02-08; First posted 2018-02-15 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-11

CONDITIONS: Hip Pain
Keywords: metal ion levels, total hip replacement, Trident II cup.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Preoperative Group (Other): This is a group of 30 patients who will be undergoing a total hip replacement with a Trident II shell. This group of patients will have their bloods drawn and tested for metal ion levels at a preoperative visit.
  Interventions: Other: Blood levels drawn
- 1 year Postoperative Group (Other): This is the same group of 30 patients who are now one year post op after having a total hip replacement with a Trident II shell. This group of patients will have their bloods drawn and tested for metal ion levels at their one year visit.
  Interventions: Other: Blood levels drawn

INTERVENTIONS:
Other: Blood levels drawn — The patients will have their bloods drawn at the Hospital for Special Surgery during their regular, standard of care visit. The laboratory at the Hospital for Special Surgery will then test their bloods to determine the metal ion levels.

SUMMARY:
Metal Ions levels of cobalt, chromium, and titanium in 40 patients preoperatively and at least 1 year status post total hip replacement with the Trident II Tritatnium system using an MDM liner and ceramic head. Are cobalt, chromium, and titanium levels in patients who undergo a total hip replacement with a Trident II Tritanium system, MDM liner, and ceramic head normal one year after surgery? Investigators expect to find normal levels of metal ions (cobalt, chromium, and titanium) after total hip replacement using Trident II Tritanium cups with an MDM liner and a ceramic head. The primary outcome (PO) is blood metal ion levels of cobalt, chromium, and titanium (concentration of metal ions in blood). Blood will be drawn in the 3rd Floor West of the Main Building, and then tested for metal ions in the Hospital for Special Surgery laboratory. The bloods will be drawn at a preoperative visit and at a one year visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will be undergoing a total hip replacement with a Stryker Trident II cup
2. Patients have signed an Institutional Review Board (IRB) approved consent form
3. Patient is 21-80
4. Patient has a diagnosis of Non-Inflammatory Degenerative Joint Disease
5. Patient is willing and able to comply with postoperative scheduled clinical evaluations.

Exclusion Criteria:

1. Patients who have not been consented as part of the Collaborative Orthopaedic Replacement Registry (CORRe) database
2. Patients with other joint replacements (shoulder/knee)
3. Patients with bilateral hip replacements
4. Prisoners
5. International Patients

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Metal Ion levels before and 1 year after a total hip replacement with a Trident II Cup | 1 year
  The primary outcome (PO) is blood metal ion levels of cobalt, chromium, and titanium (concentration of metal ions in blood). Blood will be drawn in the 3rd Floor West of the Main Building, and then tested for metal ions in the Hospital for Special Surgery laboratory.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No